CLINICAL TRIAL: NCT06455904
Title: Effects Of Concentric Cycling Training Protocol During (Neo)Adjuvant Chemotherapy in Breast Cancer Patients: PROTECT-07 Study
Acronym: PROTECT-07
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-005
Record Dates: First submitted 2024-05-30; First posted 2024-06-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an interventional, randomized controlled, prospective, multicenter and adaptive study aimed at investigating the effect of a concentric pedaling training program carried out during (neo)adjuvant chemotherapy in addition to usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): This group of patients will perform concentric cycling training program during the chemotherapy treatment.
  Interventions: Procedure: Training sessions
- Control group (No Intervention): This group of patients will benefit from standard care without additional training program.

INTERVENTIONS:
Procedure: Training sessions — The training program will be performed during 15 weeks, with one session per week.
  Arms: Training group

SUMMARY:
The association of anthracyclines (ANT) and paclitaxel (Tax) is one of the main treatments used in breast cancer. These treatments are known to induce severe side effects such as a decrease in overall exercise capacity (physical condition) in response to muscle and cardiorespiratory alterations. If exercise may be an effective preventive strategy, it seems important to prescribe the most efficient exercise modality. Among them, concentric cycling (i.e., classic cycling) can significantly induce metabolic stimulus, which is needed for maintaining exercise capacity. The PROTECT-07 study aims to demonstrate the superiority of a training program based on concentric cycling during chemotherapy compared to standard treatment. The duration of the training program is 15 weeks with one session per week.

DETAILED DESCRIPTION:
There will be two groups of patients after drawing lots using a process called randomization. The probability is one in two of being in the group participating in the training program, the other group following the standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥ 18 years old
* Stage I to III breast cancer
* Patient currently planning (neo)adjuvant treatment combining anthracycline-cyclophosphamide and weekly paclitaxel (± trastuzumab)
* Affiliation to a social security system
* Able to speak, read and understand French

Exclusion Criteria:

* No prior chemotherapy treatment
* Any known cardiac or vascular pathology
* Contraindications to physical fitness assessment
* Protected adult
* Psychiatric, musculoskeletal or neurological problems
* Pregnant or breastfeeding woman (NB: this population is already subject to a contraindication to (neo)adjuvant treatment. For women of childbearing age, a betaHCG dosage is already carried out systematically before the start of chemotherapy and information on the need for contraception throughout the chemotherapy period is provided before the start of treatment. As part of this study, only the presence of this test with a negative result at the start of chemotherapy will be checked. inclusion, if available).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2027-01-13 (Estimated); Study Completion 2027-01-13 (Estimated)

PRIMARY OUTCOMES:
Overall exercise capacity | At week 18 (the end of chemotherapy treatment)
  To investigate the superiority of a concentric pedaling training program during (neo)adjuvant chemotherapy versus the absence of a training program in patients with early breast cancer. The overall exercise capacity is assessed by the 6-minute walk test (TDM6) between the two groups.

SECONDARY OUTCOMES:
Physiological variables associated with exercise capacity - cardiorespiratory capacity | At weeks 8.
  To examine the effects of the training program on VO2max.
Physiological variables associated with exercise capacity - cardiorespiratory capacity | At week 18 (the end of chemotherapy treatment)
  To examine the effects of the training program on VO2max.
Physiological variables associated with exercise capacity - muscle function | At weeks 8.
  To examine the effects of the training program on maximal aerobic power determined as the lowest exercise intensity inducing a plateauing of O2 consumption during a maximum exercise test.
Physiological variables associated with exercise capacity - muscle function | At week 18 (the end of chemotherapy treatment)
  To examine the effects of the training program on maximal aerobic power determined as the lowest exercise intensity inducing a plateauing of O2 consumption during a maximum exercise test.
Physiological variables associated with exercise capacity - body composition | At weeks 8.
  To examine the effects of the training program on lean mass, fat mass, muscle mass assessed by bioimpedancemetry.
Physiological variables associated with exercise capacity - body composition | At week 18 (the end of chemotherapy treatment)
  To examine the effects of the training program on lean mass, fat mass, muscle mass assessed by bioimpedancemetry.
Physiological variables associated with exercise capacity - muscle architecture | At weeks 8.
  To examine the effects of the training program on muscle thickness assessed by ultrasonography.
Physiological variables associated with exercise capacity - muscle architecture | At weeks 8.
  To examine the effects of the training program on fascicle length assessed by ultrasonography.
Physiological variables associated with exercise capacity - muscle architecture | At weeks 8.
  To examine the effects of the training program on cross-sectional area assessed by ultrasonography.
Physiological variables associated with exercise capacity - muscle architecture | At week 18 (the end of chemotherapy treatment)
  To examine the effects of the training program on muscle thickness assessed by ultrasonography.
Physiological variables associated with exercise capacity - muscle architecture | At week 18 (the end of chemotherapy treatment)
  To examine the effects of the training program on fascicle length assessed by ultrasonography.
Physiological variables associated with exercise capacity - muscle architecture | At week 18 (the end of chemotherapy treatment)
  To examine the effects of the training program on cross-sectional area assessed by ultrasonography.
Psychosocial variables associated with exercise capacity - quality of life | At weeks 8.
  To examine the effects of the training program with the FACT-G questionnaire
Psychosocial variables associated with exercise capacity - quality of life | At week 18 (the end of chemotherapy treatment)
  To examine the effects of the training program with the FACT-G questionnaire
Psychosocial variables associated with exercise capacity - fatigue | At weeks 8.
  To examine the effects of the training program with the FACIT-F questionnaire
Psychosocial variables associated with exercise capacity - fatigue | At week 18 (the end of chemotherapy treatment)
  To examine the effects of the training program with the FACIT-F questionnaire
Psychosocial variables associated with exercise capacity - appetite level | At weeks 8.
  To examine the effects of the training program with the FAACT questionnaire
Psychosocial variables associated with exercise capacity - appetite level | At week 18 (the end of chemotherapy treatment)
  To examine the effects of the training program with the FAACT questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: BENDER Laura, MD, Principal Investigator — Institut de cancérologie Strasbourg Europe
Locations (2):
- France (2):
  - Hôpitaux civils de Colmar, Colmar
  - Institut de cancérologie Strasbourg Europe, Strasbourg